CLINICAL TRIAL: NCT02844153
Title: Metformin Use in Chronic Kidney Disease: The CKD-Met Study
Acronym: CKD-Met
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0408
Record Dates: First submitted 2016-07-20; First posted 2016-07-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Type 2 Diabetes; Chronic Kidney Disease
Keywords: Metformin; type 2 diabetes; chronic kidney disease; antidiabetic medications; lactic acidosis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic; Acidosis, Lactic

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 6 groups, for each CKD stage (1, 2, 3a, 3b, 4, 5): All patients with type 2 diabetes seen for the first time by a nephrologist.
  Interventions: Other: modalities of metformin prescription

INTERVENTIONS:
Other: modalities of metformin prescription — Metformin prescription or not, in each CKD stage

SUMMARY:
Metformin is the most widely prescribed oral treatment for diabetes, and the only one that showed a survival benefit.

Yet, there is no consensus on the optimal dose and withdrawal of metformin in chronic kidney disease (CKD) patients.

The aim of the study is to describe the use and side-effects of metformin in CKD patients in routine practice.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or more
* Type 2 diabetes
* Seen by a nephrologist (consultation or hospitalization) between March 2014 and March 2020 in the Department of Nephrology, Lyon Sud university hospital, France

Exclusion Criteria:

* On-going treatment by dialysis
* Kidney transplantation
* Type 1 diabetes
* Missing data (metformin treatment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with type 2 diabetes seen by a nephrologist at the University hospital of Lyon Sud, between March 2014 and March 2020
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-03; Primary Completion 2018-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients receiving metformin | every January 1st up to 2020
  metformin use during chronic kidney disease. Percentage of patients receiving metformin will be recorded.

SECONDARY OUTCOMES:
Dose of metformin | every January 1st up to 2020
  metformin use during chronic kidney disease. Dose of metformin will be recorded.
Occurence of reasons for non-prescription of metformin | every January 1st up to 2020
  metformin use during chronic kidney disease. Occurence of reasons for non-prescription of metformin will be recorded.
CKD stages | every January 1st up to 2020
  CKD stages will be recorded.
Doses of oral antidiabetes medications | every January 1st up to 2020
  Oral antidiabetic medications use during chronic kidney disease. Doses of oral antidiabetes medications (sulfonylureas, alpha-glucosidase inhibitors, Dipeptidyl peptidase-4 (DPP4) inhibitors, incretin mimetics, SGLT2 inhibitors) will be recorded.
starting time of insulin | every January 1st up to 2020
  need for insulin
occurrence of lactic acidosis | every January 1st up to 2020
  data file analysis and record of lactic acidosis episodes

CONTACTS AND LOCATIONS:
Overall Officials: Denis FOUQUE, MD PhD, Principal Investigator — Claude Bernard University, Lyon, France, Lyon Sud university hospital
Locations (1):
- Claude Bernard University, Lyon, France, Lyon Sud university hospital, Pierre-Bénite, France

REFERENCES:
- [Derived] Coliche V, Koppe L, Laville M, Nouvier M, Pelletier S, Trolliet P, Fouque D. Metformin misuse in chronic kidney disease. Diabetes Metab. 2020 Sep;46(4):337-339. doi: 10.1016/j.diabet.2018.07.005. Epub 2018 Jul 24. No abstract available. PMID 30145030